CLINICAL TRIAL: NCT03923036
Title: Anticancer Drug-induced Cardiac Adverse Events in Metastatic Colorectal Cancer: Insights From the French County Calvados Registry
Brief Title: Anticancer Vigilance Of Cardiac Events (AVOCETTE) in Metastatic Colorectal Cancer
Acronym: AVOCETTE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: TPS 68479
Record Dates: First submitted 2018-10-12; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Antineoplastic Agents; Fluorouracil; Irinotecan; Oxaliplatin; Bevacizumab; aflibercept; Capecitabine; Cetuximab; Panitumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic colorectal cancer: The French county Calvados registry of digestive cancers will allow to identify patients with a metastatic colorectal cancer diagnosed between 2004 and 2014.
  Patients will be included if the cancer was diagnosed at the metastatic stage between 2004 and 2014 or non-metastatic before 2004 that became metastatic between 2004 and 2014 (synchronous and metachronous tumors)
  Interventions: Drug: Antineoplastic Agents

INTERVENTIONS:
Drug: Antineoplastic Agents — Exposure measurement to any anticancer drug in its therapeutic use for the metastatic colorectal cancer with its posology and duration (the list provided is non-limitative). Exposure to anticancer drugs for another indication than the colorectal cancer will also be collected.
  Other Names: fluorouracile; irinotecan; oxaliplatine; bevacizumab; aflibercept; capecitabine; cetuximab; panitumumab

SUMMARY:
This study is a retrospective observational study that evaluates the rate of cardiovascular adverse events leading to hospitalization in metastatic colorectal cancer in the French county Calvados by drug exposure.

DETAILED DESCRIPTION:
This study investigates the characteristics of cardiovascular adverse events leading to hospitalization in metastatic colorectal cancer. Descriptive analysis will include incidence, type of cardiovascular adverse events.

We will explore the incidence of cardiovascular adverse events with regard of the antineoplastic drug exposures. This will provide information about the individual drug safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a metastatic colorectal cancer diagnosed between 2004 and 2014 in the French county Calvados

Exclusion Criteria:

* Minors < 18 year old
* Patients without a metastatic colorectal cancer diagnosed between 2004 and 2014 in the French county Calvados

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exhaustive population of metastatic colorectal cancers in the French county Calvados registry diagnosed between 2004 and 2014 (synchrone and metachrone diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Difference in rates of cardiovascular adverse events leading to hospitalization between chemotherapy treated patients and chemotherapy-free patients. | Between 2004 and 2017
  Any cardiovascular adverse event (e.g. the non limitative list: ischaemic heart disease, heart failure, hypertension, ischaemic stroke, embolic or thrombotic events, arrhythmias, conductive disorders) that was the primary diagnosis of a hospital admission.
  Any anticancer drug (chemotherapy) intake will be considered for the primary analysis.
  We will use a competing risk statistical model.

SECONDARY OUTCOMES:
Risk of cardiovascular adverse events (any) for each individual anticancer drug. | Between 2004 and 2017
  Drug exposure will be defined as a binary variable for each drug. (intakes/no intakes). A competing risk model will be used.
Risk of cardiovascular adverse events (any) for each anticancer drugs combination/protocol | Between 2004 and 2017
  Drugs combination will be defined as a binary variable for each protocol. (intakes/no intakes).
Risk of individual cardiovascular adverse events of chemotherapy treated patients versus chemotherapy-free patients | Between 2004 and 2017
  Several individual cardiovascular adverse events will be assessed in separate analyses: ischaemic heart disease, heart failure, hypertension, ischaemic stroke, embolic or thrombotic events, arrhythmias, conductive disorders). A competing risk model will be used
Dose-effect relation ship between individual anticancer drugs and cardiovascular adverse events | Between 2004 and 2017
  Dose will be approached by the number of cycles of the anticancer drug and by the cumulative dose (in milligram) received.
Dose-effect relation ship between individual anticancer drugs combination/protocol and cardiovascular adverse events | Between 2004 and 2017
  Dose will be approached by the number of cycles of the anticancer drugs combination/protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Alexandre, MD, PhD, Principal Investigator — CHU CAEN
Locations (1):
- CHU Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided